CLINICAL TRIAL: NCT02968901
Title: Prospective, Multicenter, Open-label Study Evaluating the Effects of First-line Oral Combination Therapy of Macitentan and Tadalafil in Patients With Newly Diagnosed Pulmonary Arterial Hypertension (OPTIMA).
Brief Title: Clinical Study Evaluating the Effects of First-line Oral cOmbination theraPy of maciTentan and tadalafIl in Patients With Newly Diagnosed pulMonary Arterial Hypertension (OPTIMA)
Acronym: OPTIMA
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AC-055-405
Record Dates: First submitted 2016-11-14; First posted 2016-11-21 (Estimated); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — macitentan; Tadalafil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- bitherapy (Experimental): Macitentan and tadalafil
  Interventions: Drug: macitentan; Drug: tadalafil

INTERVENTIONS:
Drug: macitentan — used in open label
Drug: tadalafil — used in open label

SUMMARY:
The purpose of the study is to document the effect of first line dual oral combination therapy with macitentan 10mg and tadalafil 40mg on pulmonary vascular resistance (PVR) in treatment-naïve patients with newly diagnosed pulmonary arterial hypertension (PAH).

ELIGIBILITY:
Inclusion Criteria :

1. Signed informed consent prior to any study-mandated procedure.
2. Male or female ≥ 18 and ≤ 75 years of age at screening.
3. Initial PAH diagnosis < 6 months prior to Day 1.
4. Right heart catheterization (RHC) performed between Day -28 and Day 1 (RHC data obtained at the study site within this time frame, but before the study, i.e., before signed informed consent, are acceptable), meeting all the following criteria:

   * Resting mean pulmonary arterial pressure (mPAP) ≥ 25 mmHg.
   * Pulmonary capillary wedge pressure (PCWP) or left ventricular end diastolic pressure (LVEDP) ≤ 15 mmHg.
   * PVR ≥ 400 dyn·sec/cm5 (≥ 5 Wood units) if PCWP < 12 mmHg OR PVR ≥ 500 dyn·sec/cm5 (≥ 6.25 Wood units) if PCWP in [12-15] mmHg.
   * Negative vasoreactivity test mandatory in idiopathic PAH (at this or a previous RHC).
5. World Health Organization (WHO) Functional Class (FC) II to III.
6. PAH etiology belonging to one of the following groups:

   * Idiopathic.
   * Heritable.
   * Anorexigens induced.
   * Associated with one of the following:

     * Connective tissue disease
     * Congenital heart disease with simple systemic-to-pulmonary shunt (atrial septal defect, ventricular septal defect, patent ductus arteriosus) ≥1 year after surgical repair
     * HIV infection
7. 6MWD ≥ 50 m at screening.
8. Woman of childbearing potential [see definition in Section 4.5.1] must:

   * Have a negative serum pregnancy test at the screening visit and a negative urine pregnancy test at the D1 visit, and
   * Agree to perform monthly pregnancy tests up to 30 days after EOT2, and
   * Agree to use reliable contraception [defined in Section 4.5.2] from screening up to 30 days after EOT2. Reliable contraception must be started at least 11 days prior to Day 1.

Exclusion Criteria:

1. Any PAH-specific drug therapy [e.g. any endothelin receptor antagonist, phosphodiesterase-5 inhibitors (PDE-5i), soluble guanylate cyclase stimulator, prostacyclin, prostacyclin analog, or prostacyclin receptor agonist] at any time prior to Day 1 (single-dose administration for vasoreactivity testing is permitted; previous iloprost used intermittently for the treatment of digital ulcers or Raynaud's phenomenon is permitted if stopped > 6 months prior to Day 1).
2. Subjects who changed the dose or discontinued calcium channel blockers within 1 week prior to Day 1.
3. Initiation of diuretics within 1 week prior to RCH.
4. Subjects on oral diuretics in whom the dose has not been stable for at least 1 week prior to RHC.
5. Treatment with other PDE-5i for erectile dysfunction.
6. Treatment with strong inducers of CYP3A4 (e.g., carbamazepine, rifampin, rifampicin, rifabutin, rifapentin, phenobarbital, phenytoin, and St. John's wort) ≤ 28 days prior to Day 1.
7. Treatment with strong inhibitors of CYP3A4 (e.g., ketoconazole, itraconazole, voriconazole, clarithromycin, telithromycin, nefazodone, ritonavir, boceprevir, telaprevir, saquinavir, lopinavir, fosamprenavir, darunavir, tipranavir, atazanavir, nelfinavir, amprenavir, indinavir) ≤ 28 days prior to Day 1.
8. History of priapism.
9. Significant aortic and mitral valve disease requiring a specific treatment.
10. Pericardial constriction.
11. Life-threatening arrhythmia.
12. Uncontrolled hypertension.
13. Symptomatic coronary artery disease.
14. Cardio-pulmonary rehabilitation program based on exercise (planned, or started ≤ 12 weeks prior to Day 1).
15. Body mass index (BMI) > 40 kg/m2 at screening.
16. Acute myocardial infarction ≤ 12 weeks prior to Day 1.
17. Known permanent atrial fibrillation.
18. Low blood pressure < 90/50 mmHg at screening or Day 1.
19. Ongoing or planned treatment with nitrates and/or doxazosin.
20. DLCO < 40% of predicted value (eligible only if no sign of veno-occlusive disease according to adjudication committee);
21. Presence of ≥ 1 of the following signs of relevant lung disease at any time prior to Day 1:

    * FEV1/FVC < 70% and FEV1 < 65% of predicted after bronchodilator administration;
    * Total Lung Capacity (TLC) < 60% of predicted.
22. Known or suspicion of pulmonary veno-occlusive disease (PVOD).
23. Severe renal insufficiency (estimated creatinine clearance ≤ 30 mL/min/1.73m²) assessed by central laboratory at screening.
24. Ongoing or planned dialysis.
25. Documented severe hepatic impairment (with or without cirrhosis) according to National Cancer Institute organ dysfunction working group criteria, defined as total bilirubin > 3 x ULN accompanied by AST > ULN (assessed by central laboratory at screening) and/or Child-Pugh Class C.
26. Serum AST and/or ALT > 3 x ULN (assessed by central laboratory at screening).
27. Porto-pulmonary hypertension.
28. Hemoglobin < 100 g/L assessed by central laboratory at screening.
29. Hypersensitivity to any active substance or excipient of macitentan or tadalafil formulation.
30. Loss of vision in one eye because of non-arteritic anterior ischemic optic neuropathy (NAION), regardless of whether or not this episode was in connection with previous PDE-5i exposure.
31. Hereditary degenerative retinal disorders, including retinitis pigmentosa.
32. Pregnancy, breast-feeding, intention to become pregnant during the study or woman of childbearing potential not agree to use reliable method of contraception from screening up to 30 days after EOT2.
33. Hereditary problems of galactose intolerance, Lapp lactase deficiency, glucosegalactose malabsorption.
34. Any factor or condition likely to affect protocol compliance of the patient as judged by the investigator.
35. Treatment with another investigational drug (planned, or taken ≤ 12 weeks prior to Day 1).
36. Concomitant life-threatening disease with a life expectancy < 12 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2018-09-10 (Actual); Study Completion 2018-09-10 (Actual)

PRIMARY OUTCOMES:
pulmonary vascular resistance (PVR) | 16 weeks
  Change from Baseline to Week 16 in percentage of patients with clinically meaningful improvement of PVR (decrease of 30% from baseline to Week 16)

SECONDARY OUTCOMES:
mean right atrial pressure (mRAP) | Week 16
  Change from Baseline to Week 16 in mean right atrial pressure (mRAP)
6MWD | Week 16
  Change from Baseline to Week 16 in 6MWD
level NT-proBNP | Week 16
  Change in NT-proBNP from baseline to Week 16
mean pulmonary arterial pressure (mPAP) | Week 16
  Change from Baseline to Week 16 in mean pulmonary arterial pressure (mPAP)
cardiac index (CI) | Week 16
  Change from Baseline to Week 16 in cardiac index (CI).
total pulmonary resistance (TPR) | Week 16
  Change from Baseline to Week 16 in total pulmonary resistance (TPR)
mixed venous oxygen saturation (Sv02) | Week 16
  Change from Baseline to Week 16 in mixed venous oxygen saturation (Sv02)
WHO functional class | Week 16
  Change from baseline to Week 16 in WHO functional class and Percentage of patients with improvement/worsening of WHO functional class from baseline to Week 16
Number of treatment goals | Week 16
  Number of treatment goals (score 0 or 1 per goal, i.e. total score 0-5) met at Week 16: WHO-FC I or II; Cardiac index > 2.8 L/min/m²; mRAP < 8 mmHg; 6MWD > 400 m; NT-proBNP < 3xULN

CONTACTS AND LOCATIONS:
Locations (18):
- France (18):
  - Hôpital Jean Minjoz, Besançon
  - Hôpital de Haut Levêque, Bordeaux
  - Hôpital Côte de Nacre, Caen
  - CHU Site du Bocage, Dijon
  - Hôpital Albert Michallon, Grenoble
  - Hôpital Bicètre, Le Kremlin-Bicêtre
  - Hôpital Dupuytren, Limoges
  - Hôpital Louis Pradel, Lyon
  - Hôpital Timone Adultes, Marseille
  - Hôpital Arnaud de Villeneuve, Montpellier
  - CHR La Miletrie, Poitiers
  - Hôpital Robert Debré, Reims
  - Hôpital Pontchaillou, Rennes
  - Hôpital Charles Nicolle, Rouen
  - Hôpital Nord, Saint-Priest-en-Jarez
  - Hôpital Civil, Strasbourg
  - Hôpital Larrey, Toulouse
  - Hôpital Bretonneau, Tours

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Clinical study evaluating the effects of first-line oral combination therapy of macitentan and tadalafil in patients with newly diagnosed pulmonary arterial hypertension (OPTIMA) — https://www.clinicaltrialsregister.eu/ctr-search/trial/2015-002078-19/results